CLINICAL TRIAL: NCT01414959
Title: Target Site Pharmacokinetics of Doripenem at Steady State in Intubated Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Zeitlinger, Professor Dr., Medical University of Vienna
Other Study IDs: Dori_MD_ICU
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Pneumonia; Abdominal Infection; Urinary Tract Infection
Keywords: intensive care patient; intubation; (please change wording as you like!)
MeSH Terms: conditions — Pneumonia; Intraabdominal Infections; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma broncheoalvoeolar lavage microdialysates
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will measure the pharmacokinetics of doripenem in skeletal muscle, subcutaneous adipose tissue, bronchoalveolar lavage and plasma of intubated intensive care patients.

DETAILED DESCRIPTION:
Methods: microdialysis, blood sampling, bronchoalveolar lavage

ELIGIBILITY:
Inclusion Criteria:

* endotracheal intubation; pneumonia or complicated abdominal infection or complicated urinary tract infection

Exclusion Criteria:

* allergy to doripenem, hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intubated patients, intensive care
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zeitlinger, MD, Principal Investigator — Medical Universit of Vienna
Locations (1):
- Med. Univ. of Vienna, Vienna, Austria